CLINICAL TRIAL: NCT06696209
Title: Analysis of Withdrawal Time in Upper Gastrointestinal Endoscopy as Procedure Time: a Randomised, Parallel, Double-blinded, Multicenter, International Clinical Trial
Brief Title: To Evaluate the Best Metric for Inspection Time During a Diagnostic and/or Surveillance Upper Gastrointestinal Endoscopy (Age ≥ 18 Years, Informed Consent), Between Total Inspection Time Versus Withdrawal Time, for the Identification of Malignant Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Maria Inês Viegas, Medical Doctor, Portuguese Oncology Institute, Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PortugueseOIC 006
Record Dates: First submitted 2024-10-30; First posted 2024-11-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Premalignant Conditions; Malignant Lesions; Gastric; Esophageal; Duodenal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analysis of the withdrawal time of the Upper Gastrointestinal Endoscopy (Active Comparator)
  Interventions: Other: Analysis of the withdrawal time of the Upper Gastrointestinal Endoscopy; Other: Upper gastrointestinal endoscopy: Common Practices
- Analysis of the total time of the Upper Gastrointestinal Endoscopy (Active Comparator)
  Interventions: Other: Analysis of the total time of the Upper Gastrointestinal Endoscopy; Other: Upper gastrointestinal endoscopy: Common Practices

INTERVENTIONS:
Other: Analysis of the withdrawal time of the Upper Gastrointestinal Endoscopy — Time of last esophageal image - time of first image of the second portion of the duodenum.
  Arms: Analysis of the withdrawal time of the Upper Gastrointestinal Endoscopy
Other: Analysis of the total time of the Upper Gastrointestinal Endoscopy — Time of last esophageal image - time of first esophageal image
  Arms: Analysis of the total time of the Upper Gastrointestinal Endoscopy
Other: Upper gastrointestinal endoscopy: Common Practices — Execution of UGE using high-resolution endoscopes, with the option of virtual chromoendoscopy, according with the physician's preference. Possible optimization of visualization with washing and/or the use of simethicone or similar, as pre-medication or during the examination, according with the physician's preference. Patients will be randomised to one of the following measurements-total time versus withdrawal time-in a parallel 1:1 scheme.
  The allocation of the randomisation group will be computer-generated. The endoscopist must record the time at which the following three anatomical structures are reached (either by noting during the procedure or based on the information in the photographic documentation), before any biopsies or therapeutic interventions, in the format xxh:xxmin:xxsec:
  1. First esophageal image;
  2. First image of the second portion of the duodenum;
  3. Last esophageal image.

SUMMARY:
Gastric cancer is the fifth cause of cancer-related mortality worldwide. Gastric carcinogenesis involves the progression from premalignant conditions such as atrophic gastritis and intestinal metaplasia to premalignant lesions like dysplasia, and ultimately carcinoma. Most diagnoses of gastric cancer are made at advanced stages, with a five-year relative survival rate of 36%. Therefore, early detection of premalignant conditions and lesions is crucial, as it allows for timely surveillance and treatment, which can improve patient survival.

Upper gastrointestinal endoscopy (UGE) is the first-line examination for diagnosing upper gastrointestinal tract pathology, particularly oncological conditions. The European Society of Gastrointestinal Endoscopy (ESGE) and the United European Gastroenterology (UEG) have established that UGE quality is a priority, identifying specific quality parameters, such as the duration of the procedure, which is the most extensively studied parameter.

According to ESGE recommendations, all UGE reports should include the procedure time (goal: ≥90% of reports), which should be seven minutes or longer for surveillance of intestinal metaplasia. This time threshold follows a study that established a causal relationship between longer procedures (≥ seven minutes) and a higher detection rate of premalignant gastric conditions and lesions. Subsequent observational studies have generally shown that setting a minimum procedure time increases the detection rate of lesions.

The definition of procedure time varies between studies, being described as the time from intubation to extubation, but also as the time for withdrawing the endoscope from the second portion of the duodenum (D2) to extubation, also known as withdrawal time.

The hypothesis under study is that a better definition of the most appropriate time for a diagnostic UGE could standardize reports, improve malignant lesion detection rates, and reduce the rate of undiagnosed cancers, without any additional risk to patients.

Existing studies have been retrospective or comparative between different temporal cohorts, with no prospective or randomised comparative studies, nor any studies comparing the two existing metrics. Therefore, the aim of this study is to evaluate the best metric for inspection time during a diagnostic and/or surveillance UGE, between total inspection time versus withdrawal time, for the identification of malignant lesions.

DETAILED DESCRIPTION:
Execution of UGE using high-resolution endoscopes, with the option of virtual chromoendoscopy, according with the physician's preference. Possible optimization of visualization with washing and/or the use of simethicone or similar, as pre-medication or during the examination, according with the physician's preference. Patients will be randomised to one of the following measurements-total time versus withdrawal time-in a parallel 1:1 scheme. The allocation of the randomisation group will be computer-generated. The endoscopist must record the time at which the following three anatomical structures are reached (either by noting during the procedure or based on the information in the photographic documentation), before any biopsies or therapeutic interventions, in the format xxh:xxmin:xxsec:

1. First esophageal image;
2. First image of the second portion of the duodenum;
3. Last esophageal image.

The endoscopist will perform the UGE for as long as clinically necessary, which may be shortened if there is any need to interrupt the procedure for any clinical reason (such as intolerance or other), without any minimum or maximum time limits.

Although this is a non-interventional study that does not involve any modification to daily clinical practice, regarding the analyzed UGE, the study will be submitted for evaluation by the Ethics Committee of the Portuguese Institute of Oncology of Coimbra and will be performed in accordance with the principles of the Helsinki Declaration. All analyzed data will be kept confidential, and the investigators will ensure the anonymity of the patients included during data analysis and publication.

This study aims to define the best metric for quantifying the most appropriate time for performing a diagnostic or surveillance UGE. To our knowledge, all existing studies on the topic of procedure time in UGE are observational. This study will be the first randomised clinical trial in this area, with the purpose of providing a systematic evaluation that will contribute to the optimization of quality measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnostic or surveillance upper gastrointestinal endoscopy for premalignant conditions
* Informed consent for the execution of the upper gastrointestinal endoscopy and participation in the study

Exclusion Criteria:

* Previous esophagus, stomach, or duodenum surgery
* Known or suspected neoplasia
* Therapeutic procedure (polypectomy, argon plasma coagulation, hemostasis, others)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1290 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Detection rate of premalignant conditions and malignant lesions, defined as the total number of lesions in the esophagus, stomach, or duodenum detected per randomisation group, confirmed by histological evaluation (if necessary) | One month

SECONDARY OUTCOMES:
• Complications: related to sedation, cardiopulmonary adverse events, bleeding, perforation, others. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Portuguese Institute of Oncology, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes